CLINICAL TRIAL: NCT00088803
Title: The Incidence, Inheritance, and Prognostic Significance of Polymorphisms in the RASSF1A Gene in Children With Wilms Tumors
Brief Title: DNA Variations in the Gene in Young Patients With Wilms' Tumor
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AREN04B1; COG-AREN04B1 (Other: Children's Oncology Group); UTSMC-0390080; CDR0000366933 (Other: Clinical Trials.gov); NCI-2009-00417 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Kidney Cancer
Keywords: recurrent Wilms tumor and other childhood kidney tumors; stage I Wilms tumor; stage II Wilms tumor; stage III Wilms tumor; stage IV Wilms tumor; stage V Wilms tumor
MeSH Terms: conditions — Kidney Neoplasms; Wilms Tumor | interventions — Genetic Testing; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: molecular genetic technique
Genetic: polymerase chain reaction
Genetic: polymorphism analysis

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at DNA variations in the RASSF1A gene in young patients with Wilms' tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the presence of the A133S polymorphism in the RASSF1A tumor suppressor gene by screening germline DNAs of children with Wilms' tumor.
* Determine the inheritance pattern of the A133S polymorphism by evaluating the parents of children who carry this polymorphism.

Secondary

* Determine the differences in age at diagnosis, stage, histology, site of primary tumor, and outcome, between patients with vs without the A133S polymorphism.
* Determine whether the S131F RASSF1A variant is a true polymorphism in these patients.
* Determine the polymorphic differences in this gene between these patients based on ethnicity and sex.

OUTLINE: This is a multicenter study. Patients are stratified according to age at diagnosis, stage, histology, site of primary tumor, and outcome.

Genomic DNA samples are purified from peripheral blood of patients and controls and analyzed by polymerase chain reaction for the RASSF1A gene. DNA is also analyzed from parents of patients with the A133S polymorphism.

PROJECTED ACCRUAL: A total of 471 participants (229 Wilms' tumor patients and 200 control participants plus 42 parents) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Wilms' tumor OR
* Control participants matched for race, sex, and age

  * No prior or concurrent history of cancer OR
* Parents of children involved in the study

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Diagnosis of Wilms' tumor or control participants matched for race, sex, and age.
Sampling Method: Non-Probability Sample
Enrollment: 471 (Estimated)
Dates: Start 2004-08; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Presence of the A133S polymorphism of the RASSF1A tumor suppressor gene in germline DNAs of children with Wilms' tumor
Inheritance pattern of the A133S polymorphism in the parents of children who carry this polymorphism

SECONDARY OUTCOMES:
Differences in age at diagnosis, stage, histology, site of primary tumor, and outcome between patients with vs without the A133S polymorphism
Whether the S131F RASSF1A variant is a true polymorphism
Polymorphic differences in this gene based on ethnicity and sex

CONTACTS AND LOCATIONS:
Overall Officials: Gail E. Tomlinson, MD, PhD, Study Chair — Simmons Cancer Center
Locations (232):
- United States (205):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of South Alabama Cancer Research Institute, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - Children's Hospital and Health Center, San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital of Denver, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - University of Connecticut Comprehensive Cancer Center at University of Connecticut Health Center, Farmington, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Shands Cancer Center at the University of Florida Health Science Center, Gainesville, Florida
  - Joe DiMaggio Children's Hospital at Memorial, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic-Orlando, Orlando, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Mountain States Tumor Institute - Boise, Boise, Idaho
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Medical Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - St. Vincent Hospitals and Health Care Centers, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Walter Reed Army Medical Center, Silver Spring, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Baystate Regional Cancer Program at Baystate Medical Center, Springfield, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health and DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Children's Hospitals and Clinics - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Hospitals and Clinics - Minnesota, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Omaha, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey at Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Valerie Fund Children's Center at Atlantic Health, Summit, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Comprehensive Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospitals, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Center of University Health Systems of Eastern Carolina, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Dakota Cancer Institute at Innovis Health - Dakota Clinic, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Forum Health-Tod Childrens Hospital, Youngstown, Ohio
  - Children's Hospital at Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Doernbecher Children's Hospital at Oregon Health & Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sioux Valley Hospital at University of South Dakota Medical Center, Sioux Falls, South Dakota
  - East Tennessee State University Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MBCCOP - South Texas Pediatrics, San Antonio, Texas
  - Methodist Cancer Center at Methodist Specialty and Transplant Hospital, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Center for Cancer Prevention and Care at Scott and White Clinic, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Carilion Medical Center for Children, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Cabell Huntington Hospital, Huntington, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (5):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre de Recherche du Centre Hospitalier de l'Universite Laval, Sainte-Foy, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- Starship Children's Health, Auckland, New Zealand
- Puerto Rico (2):
  - Puerto Rico Cancer Center at University of Puerto Rico - Medical Sciences Campus, San Juan
  - San Jorge Childrens Hospital, Santurce
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne